CLINICAL TRIAL: NCT05565313
Title: Predicting Radiological Extranodal Extension in Oropharyngeal Carcinoma Patients Using AI
Acronym: AI4rENE
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Brigham and Women's Hospital (Other); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: W 22 03 00000 - P0471 V1.2
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Development and validation of a model that predicts rENE from radiological imaging using annotated / labeled scans by means of deep learning

DETAILED DESCRIPTION:
Oropharyngeal squamous cell carcinoma (OPSCC) is a rare cancer (incidence ~700 per year in the Netherlands), originating in the middle part of the throat. In OPSCC, nodal status is an important prognostic factor for survival. In the clinical TNM (tumor node metastases) system, nodal status is mainly defined by the size, number and laterality of nodal metastases. In surgically treated patients the pathological TNM classification includes the presence of pathological extranodal extension (pENE). pENE is a predictor for poor outcome and also an indication for the addition of chemotherapy to postoperative radiation. However, most patients with OPSCC are treated non-surgically by means of radiation or chemoradiation and thus information about pENE is lacking. Recently, extranodal extension on diagnostic imaging has been associated with prognosis in OPSCC patients. It is anticipated that in the near future radiological ENE (rENE) may be included in the cTNM classification system for refinement of outcome prediction in patients with nodal disease. The diagnosis of rENE on radiological imaging is new and not trivial and we hypothesize that Artificial Intelligence (AI) may support the radiologist in detecting rENE. In this study we aim to develop and validate a model that predicts rENE from radiological imaging using annotated / labeled scans by means of deep learning

ELIGIBILITY:
Inclusion criteria:

* Non-metastatic (M0) node-positive HPV+ and HPV- oropharyngeal carcinoma
* Treated between 2008 to 2019
* Curative intent
* Radiation only or concurrent chemoradiation
* Modern treatment modality: IMRT / VMAT
* diagnostic/staging image scanning protocols available (contrast-enhanced CT with 2-3 mm slice thickness and/or MR with 3 mm slice thickness)

Exclusion criteria:

* removal of lymph node (LN) (excisional biopsy or neck dissection [ND]) prior to staging CT/MR scan
* no available imaging within 2 months prior to radiotherapy (RT)"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria:
  * Non-metastatic (M0) node-positive HPV+ and HPV- (human papilloma virus) oropharyngeal carcinoma
  * Treated between 2008 to 2019
  * Curative intent
  * Radiation only or concurrent chemoradiation
  * Modern treatment modality: IMRT / VMAT (Intensity Modulated RadioTherapy / Volumetric-Modulated Arc Therapy)
  * diagnostic/staging image scanning protocols available (contrast-enhanced CT with 2-3 mm slice thickness and/or MR (magnetic resonance) with 3 mm slice thickness)
  Exclusion criteria:
  * removal of lymph node (LN) (excisional biopsy or neck dissection [ND]) prior to staging CT/MR scan
  * no available imaging within 2 months prior to radiotherapy (RT)"
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of rENE as labeled by the radiologist, using the AI model | Baseline
  The performance of the model will be evaluated in terms of discrimination through the Harrell's C-index and the area (AUC) under the receiver operator curve (ROC) in predicting rENE.

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Percentage of people who are alive five years after their diagnosis.
Disease Free Survival | 5 years
  Percentage of people whp who are disease free five years after their diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hoebers, PhD, Principal Investigator — Maastro
Locations (3):
- Harvard Medical School and clinical faculty at Dana-Farber Cancer Institute/Brigham and Women's Hospital, Boston, Massachusetts, United States
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Maastro, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all IPD (individual participant data) underlying the results
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Starting 6 months after publication